CLINICAL TRIAL: NCT00891345
Title: A Prospective, Open Phase I Study to Investigate the Tolerability and Efficacy of Administering ALECSAT to Prostate Cancer Patients - a First Dose in Man Study
Brief Title: Safety Study of a Cytotoxic Lymphocytes (CTL) Based Prostate Cancer Therapy
Acronym: ALECSAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CytoVac A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV001
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Hormone-refractory Prostate Cancer
Keywords: hormone-refractory prostate cancer; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: ALECSAT — Autologous activated CTL and NK-cells injected as a single intravenous injection.

SUMMARY:
This study is a phase I study of a new cell based prostate cancer therapy (ALECSAT). In this therapy specific cells from the patient's own immune system are isolated, activated and re-administered to the patient to boost a specific immune response against the cancer cells. The aim of the study is to show safety and tolerability for this type of therapy. It is the hypothesis that the cells administered during the therapy will attack the tumour cells and in this way stop or slow down the progression of disease.

DETAILED DESCRIPTION:
This study is a prospective open phase I study to investigate the safety and tolerability of administration of a single dose of a cell based medicinal product (CBMP) ALECSAT.

ALECSAT is an autologous CBMP that is made from the patient's own blood cells. ALECSAT contains a large amount of tumour specific cytotoxic Lymphocytes (CTL) and Natural Killer (NK) cells that are isolated activated and amplified in number.

The CBMP is given as a slow i. v. injection to patients with prostate cancer. The patients are in the late stage of the disease where they have received hormone treatment but their disease is progressing.

The primary objective of the study is to observe if any side effects or tolerability issues occur as a consequence of the cell administration, secondarily it will be observed if any positive anti tumour effect may be observed. The study has the purpose to investigate whether treatment with ALECSAT in any way is toxic.

Trial Design: The study is an open, prospective phase I safety study of ALECSAT in prostate cancer patients.

A group consisting of 6 patients will be treated with ALECSAT according to the protocol. Then an interim analysis will be done. If there are no signs of significant toxicity related to the treatment, the study will continue with 8 more patients that will be included and treated with ALECSAT according to the phase I protocol. Thus this study will include a total of 14 patients.

The patients will after a single administration of ALECSAT be hospitalised for 3 days and will furthermore be followed closely for 7 weeks by 5 planned study visits, by the investigators at Urologisk Klinik at Fredrikssund Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Hormone-refractory prostate cancer patients
* Three consecutive rises of PSA min. 2 weeks apart, resulting in at least two 50% increases over the PSA nadir.
* Antiandrogen withdrawal for at least 4 weeks, or
* PSA progression despite secondary hormonal manipulations, or
* Progression of osseous or soft tissue lesions.
* Serum castration levels of testosterone.
* Be capable of understanding the information and giving informed consent.
* Expected survival time (life expectancy) of over 4 months.
* Adequate performance status (WHO / ECOG Performance status score 2 or less).

Exclusion Criteria:

* Patients with a low blood count (haemoglobin < 6.0 mmol/l).
* Patients with lymphocyte-numbers below 0.8.
* Patients known to be HIV and/or hepatitis positive i.e. patients positive in tests for anti-HIV-1/2; HBsAg, anti-HBc and Anti-HCV.
* Patients known to have syphilis i.e. being positive in a Treponema Pallidum test.
* Patients with uncontrolled serious bacterial, viral, fungal or parasitic infection.
* Patients must have no clinically significant autoimmune disorders or conditions of immune suppression.
* Patients that have been treated with corticosteroids (steroid hormones) or bisphosphonates or have been in chemotherapy or radiation treatment one month prior to inclusion in the clinical trial.
* Fertile patients.
* Patients that have received blood transfusions within 48 hours prior to donation of blood for ALECSAT production.
* Patients must not have been included in other clinical trials 6 weeks prior to inclusion in the trial or be enrolled in other clinical trials during the ALECSAT clinical trial.
* Any medical condition that will render participation in the study risky or, according to the investigator in charge, will make the assessment of side-effects difficult.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to show safety and tolerability for the administration of ALECSAT to enable further clinical development of the ALECSAT therapy. | Within 7 weeks

SECONDARY OUTCOMES:
The secondary endpoint for this study is to establish if any indications of a positive therapeutic effect on the prostate cancer may be observed. | Within 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Henrik Meyhoff, MD, Principal Investigator — Urologisk Klinik, Frederikssund Hospital, Frederikssundsvej 30, 3600 Frederikssund
Locations (1):
- Urological Clinic, Frederikssunds Hospital, Frederikssund, Denmark

REFERENCES:
- [Derived] Gammelgaard OL, Ehmsen S, Jylling AMB, Sandberg L, Kirkin AF, Kodahl AR, Ditzel HJ. Adoptive cell transfer therapy with ex vivo primed peripheral lymphocytes in combination with chemotherapy in locally advanced or metastatic triple-negative breast cancer: the ImmunoBreast phase Ib clinical trial. J Immunother Cancer. 2025 Dec 4;13(12):e012213. doi: 10.1136/jitc-2025-012213. PMID 41344991